CLINICAL TRIAL: NCT02097420
Title: HALO Clinical Study: A Single Arm, Prospective, Non-randomized, Multi Center Investigation of the SJM™ Masters HP™ 15mm Rotatable Mechanical Heart Valve
Brief Title: HALO: A Single Arm Prospective Investigation of the SJM™ Masters HP™ 15mm Rotatable Mechanical Heart Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL06404
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Mitral Valve Disease; Damaged Mitral Valve; Malfunctioning Mitral Heart Valve; Mitral Valve Replacement
Keywords: Mitral valve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single device arm (Other): Mitral valve replacement
  Interventions: Device: Mitral valve replacement SJM™ Masters HP™ 15mm Rotatable Mechanical Heart Valve

INTERVENTIONS:
Device: Mitral valve replacement SJM™ Masters HP™ 15mm Rotatable Mechanical Heart Valve — Implantation of the SJM™ Masters HP™ 15mm Rotatable Mechanical Heart Valve in the mitral and aortic positions

SUMMARY:
The purpose of the study is to provide evidence of safety and effectiveness of the study valve. The rationale is to offer a replacement mitral valve for patients with anatomy that is too small for the currently commercially available valves ranging in size from 16mm to 37mm.

20 subjects were enrolled as part of the IDE cohort and an additional 3 were enrolled under continued access.

DETAILED DESCRIPTION:
The study is a single arm, prospective, non-randomized, multi-center clinical investigation.

The objective of this study is to evaluate the safety and effectiveness of the 15mm MHV in subjects five years or less of age with a diseased, damaged, or malfunctioning mitral heart valve. The objective will be evaluated by assessing valve-related adverse events, subject survival, subject growth, and echocardiogram assessment of hemodynamic function through the five year follow-up visit as long as the valve remains implanted.

ELIGIBILITY:
IDE Cohort -

Inclusion Criteria:

1. Subject requires mitral valve replacement.*
2. Subject's legally authorized representative gives written consent to participate in the clinical study.
3. Subject is willing and able to return for data collection and follow-up for the duration of the clinical study.

   * Subjects undergoing concomitant procedures (e.g. valve repair) are eligible for this study other than those noted in the exclusion criteria.

Exclusion Criteria:

1. 1. Subject is > 5 years of age.
2. Subject has a contraindication to anticoagulant/antiplatelet medication.
3. Subject has a prosthetic valve(s) at a site other than the mitral valve prior to the study procedure.*
4. Subject requires concomitant replacement of the tricuspid, pulmonary, or aortic valve.
5. Subject has active endocarditis.
6. Subject has active myocarditis.
7. Subject has had an acute preoperative neurological deficit that has not returned to baseline or stabilized ≥ 30 days prior to the study procedure.
8. Subject has had an acute cardiac adverse event that has not returned to baseline or stabilized ≥48 hours prior to the study procedure.
9. Subject has a non-cardiac illness resulting in a life expectancy of < 1 year.
10. Subject has a known requirement for additional cardiac surgery within 12 months after the study procedure.
11. Subject has been previously enrolled and implanted in this study.
12. Subject is participating in another study for an investigational drug and/or device.
13. Subject has any other medical condition that in the opinion of the Investigator will interfere with the study results.

    * Subjects who have undergone a previous Ross procedure of the pulmonary valve are eligible for this study.

Continued Access Cohort-

Prospective Inclusion Criteria:

1. Subject requires mitral valve replacement.*
2. Subject's legally authorized representative gives written consent to participate in the clinical study.
3. Subject is willing and able to return for data collection and follow-up for the duration of the clinical study.

   * Subjects undergoing concomitant procedures (e.g. valve repair) are eligible for this study.

Prospective Exclusion Criteria:

1. Subject is > 5 years of age.
2. Subject has a contraindication to anticoagulant/antiplatelet medication.

Retrospective Eligibility Criteria:

1. The subject must have been ≤ 5 years of age at the time of mitral valve replacement with the 15mm MHV.
2. An implant was attempted with the 15mm MHV, where implant attempt is defined as the device physically contacting the subject's cardiac anatomy.
3. The legally authorized representative signs the study informed consent for this protocol allowing access to all relevant historical medical information and prospective follow-up (if applicable).
4. Either

   1. the legally authorized representative and site agree to follow the subject per the assessment schedule and complete all required assessments per this protocol from the time of consent going forward.

      OR
   2. the subject's status is deceased or explanted, but an implant with 15mm MHV was attempted.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2023-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles (USC), Los Angeles, California
  - University of California - Davis Medical Center, Sacramento, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - University of Missouri-Kansas City School of Medicine, Kansas City, Missouri
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - New York Presbyterian Hospital/Columbia University, New York, New York
  - Levine Children's Hospital / Sanger Heart & Vascular Institute, Charlotte, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 23 subjects were enrolled at 15 investigational sites. Twenty (20) subjects were enrolled at 14 sites in the IDE cohort. Following completion of enrollment in the IDE cohort, 3 subjects were enrolled at 3 sites in the CAP cohort. All subjects enrolled in the study were followed for up to 5 years post-implant, or until the valve was retired/explanted, whichever occurred first. Enrollment was completed in the IDE cohort on 03 March 2017 and in the CAP cohort on 12 January 2018.
Groups:
- Single Device Arm: Mitral Valve Replacement: Subjects who underwent mitral valve implantation or replacement using SJM™ Masters HP™ 15mm Rotatable Mechanical Heart Valve in the mitral and aortic positions
Period: Overall Study
Arm/Group | Single Device Arm: Mitral Valve Replacement
Started | 23
Completed | 3
Not Completed | 20
Not completed — Death | 6
Not completed — Valve explanted | 13
Not completed — Other Reason | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Device Arm: Mitral Valve Replacement
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
Weight [Mean (Standard Deviation); unit: kilograms] | 5.5 (1.9)
Height [Mean (Standard Deviation); unit: centimeters] | 60.5 (9.2)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: meter square] | 0.3 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint: Kaplan-Meier Percentage of Participants Who Remained Alive or Had Valve Explanted Due to Anatomical Growth
Description: The Kaplan-Meier method is a statistical method that summarizes the rate at which subjects survive or are free from a specified event. The method uses whether or not a subject had the specified event and their time to the specified event or the end of their follow-up to calculate the rate.
  Kaplan-Meier event rates with 95% confidence intervals would be calculated for overall survival. All follow-up time through 365 days post implant would be considered. If a subject discontinues prior to one year post implant, all available data would be included.
Time Frame: 12 months
Population: The analysis population included the subjects who were available at the time of evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Device Arm: Mitral Valve Replacement
Number analyzed (Participants) | 23
percentage of participants | 71.0 [46.3 to 85.9]

2. Primary Outcome: Primary Effectiveness Endpoint: Peak Gradient as Assessed by Echocardiography
Description: Peak gradient as assessed by echocardiography at 12 months post implant or when the valve is removed/replaced due to anatomical growth of the subject, whichever occurs first.
Time Frame: 12 months
Population: The analysis population included the 14 subjects who have completed the 12-month follow-up visit or until the valve was removed/replaced due to anatomical growth, whichever occurred first.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Device Arm: Mitral Valve Replacement
Number analyzed (Participants) | 14
mmHg | 19.8 (7.6)

3. Primary Outcome: Primary Effectiveness Endpoint: Mean Gradient as Assessed by Echocardiography
Description: Mean gradient as assessed by echocardiography at 12 months post implant or when the valve is removed/replaced due to anatomical growth of the subject, whichever occurs first.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Device Arm: Mitral Valve Replacement
Number analyzed (Participants) | 14
mmHg | 7.9 (4.6)

4. Primary Outcome: Primary Effectiveness Endpoint: Number of Participants With Valvular Regurgitation
Description: Valvular regurgitation as assessed by echocardiography at 12 months post implant or when the valve is removed/replaced due to anatomical growth of the subject, whichever occurs first.
Time Frame: 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Single Device Arm: Mitral Valve Replacement
Number analyzed (Participants) | 14
Participants
  None | 9
  Trivial | 3
  Mild (1+) | 1
  Moderate (2+) | 1
  Moderately Severe (3+) | 0
  Severe (4+) | 0
  Present/Unknown | 0
  Unknown | 0

5. Primary Outcome: Primary Safety Endpoint: Rate of Total Valve-related Adverse Events
Description: Kaplan-Meier event rates with 95% confidence intervals would be calculated for valve-related adverse events. All follow-up time through 365 days post implant would be considered. If a subject discontinues prior to one year post implant, all available data would be included.
Time Frame: 12 months
Population: The analysis population included the subjects who were available at the time of evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Device Arm: Mitral Valve Replacement
Number analyzed (Participants) | 23
percentage of participants | 64.3 [39.0 to 81.3]

6. Secondary Outcome: Percentage Change in Height Percentiles From Baseline to 12 Months
Description: Percentiles would be summarized by visit interval from baseline to 12 months for all available data. Summary statistics including number of subjects, mean and standard deviation are provided at the 12-month visit.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Single Device Arm: Mitral Valve Replacement
Number analyzed (Participants) | 14
Percentage of change | 59.4 (233.0)

7. Secondary Outcome: Percentage Change in Weight Percentiles From Baseline to 12 Months
Description: Percentiles would be summarized by visit interval from baseline to 12 months for all available data.Summary statistics including number of subjects, mean, standard deviation, and difference between visits were used for this endpoint.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Single Device Arm: Mitral Valve Replacement
Number analyzed (Participants) | 14
Percentage of change | 370.8 (812.3)

ADVERSE EVENTS:
Time Frame: 60 months
Arm/Group | Single Device Arm: Mitral Valve Replacement
All-Cause Mortality (participants affected / at risk) | 6/23
Serious Adverse Events (participants affected / at risk) | 19/23
Other Adverse Events (participants affected / at risk) | 11/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Device Arm: Mitral Valve Replacement (N=23)
Abnormal Coagulation Parameter (Blood and lymphatic system disorders) | 2
Anemias (Blood and lymphatic system disorders) | 2
Hemolysis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Atrial Tachycardia (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Heart Block (Cardiac disorders) | 2
Heart Failure (Cardiac disorders) | 1
LVOT Resection with Resection of Subaortic Membrane Myotomy (Cardiac disorders) | 1
Left Ventricle Outflow Tract Observation w/ Subaortic Obstruction (Cardiac disorders) | 1
Left Ventricular Failure (Cardiac disorders) | 1
Mitral Valve Stenosis (Cardiac disorders) | 1
Moderate Left Ventricular (LV) Dysfunction (Cardiac disorders) | 1
Pseudoaneurysm on Left Ventricular Free Wall (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Third Degree Heart Block (Complete Heart Block) (Cardiac disorders) | 3
Multiple Organ Failure (General disorders) | 1
Other (General disorders) | 4
Perivalvular Leak (General disorders) | 1 — Valve related adverse event
Bacterial Infections (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Common Cold/Upper Respiratory Tract Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic Shock Related to Presumed Pneumotosis/Nec (Infections and infestations) | 1
Viral Syndrome (Infections and infestations) | 1
Abnormal Chest X-Ray (Investigations) | 1
Abnormal Lab Value (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypervolemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Respiratory Acidosis (Metabolism and nutrition disorders) | 1
Generalized Tonic-Clonic Seizures (Nervous system disorders) | 1
Prosthetic Mitral Valve Dysfunction (Product Issues) | 1
Thrombus (Product Issues) | 2
Thrombus on Device (Product Issues) | 3 — Valve related adverse event
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2
G-Tube Procedure (Surgical and medical procedures) | 1
Acute Subdural Hematoma (Vascular disorders) | 1 — Valve related adverse event
Bleeding (Vascular disorders) | 1 — Valve related adverse event
Epistaxis (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1
Intracerebral Haemorrhage (Vascular disorders) | 1 — Valve related adverse event
Intraparenchymal Haemorrhage (Vascular disorders) | 1 — Valve related adverse event
Subdural Haemorrhage (Vascular disorders) | 1 — Valve related adverse event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Device Arm: Mitral Valve Replacement (N=23)
Abnormal Coagulation Parameter (Blood and lymphatic system disorders) | 1
Anemias (Blood and lymphatic system disorders) | 2
Hemolysis (Blood and lymphatic system disorders) | 1
Atrial Tachycardia (Cardiac disorders) | 2
Augmentation of Ascending Aorta with Pulmonary Homograft (Cardiac disorders) | 1
Elevated RV Pressure and Pulmonary Vasculature Resistance (Cardiac disorders) | 1
Infective/Bacterial Endocarditis (Cardiac disorders) | 1
Junctional Escape Rhythm/Intermittent Junctional Rhythm (Cardiac disorders) | 1
LVOT Resection (Cardiac disorders) | 1
Mitral Valve Stenosis (Cardiac disorders) | 1
Progressive LVOT Obstruction (Cardiac disorders) | 1
ST Segment Changes (Cardiac disorders) | 1
Sinus Node Dysfunction (Cardiac disorders) | 1
Third Degree Heart Block (Complete Heart Block) (Cardiac disorders) | 1
Valve Stenosis (Cardiac disorders) | 1
Fever (General disorders) | 2
Other (General disorders) | 5
Common Cold/Upper Respiratory Tract Infection (Infections and infestations) | 1
Abnormal Lab Value (Investigations) | 1
Elevated ALT Levels (Investigations) | 1
Elevated AST Levels (Investigations) | 1
Elevated Plasma Free Hemoglobin (Investigations) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Elective Procedure (Surgical and medical procedures) | 1
Elective Surgery (Surgical and medical procedures) | 1
Reoperation for Subaortic Stenosis (Surgical and medical procedures) | 1
Bleeding (Vascular disorders) | 1
Cardiogenic Shock (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT02097420/Prot_SAP_001.pdf